CLINICAL TRIAL: NCT01537341
Title: Asymmetric Locomotor Training in the Elderly to Restore Physical Function
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding was not received for this study.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UF_IOA_Pepper_Nocera
Record Dates: First submitted 2012-02-14; First posted 2012-02-23 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Disability

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional Treadmill (Active Comparator): Participants will follow the same guidelines as the split belt component but will complete the intervention on a traditional, single belt/speed treadmill.
  Interventions: Behavioral: Traditional Treadmill
- Split-belt (Experimental): Participants will walk on a custom-built split-belt treadmill comprised of two separate belts, each with its own motor, that permitted the speed of each belt (i.e. each leg) to be controlled independently.
  Interventions: Behavioral: Split-belt

INTERVENTIONS:
Behavioral: Traditional Treadmill — Participants will complete the intervention in 12-weeks, 3 times per week sessions.
  Other Names: Traditional Treadmill is a single belt/speed treadmill.
  Arms: Traditional Treadmill
Behavioral: Split-belt — Participants will complete the intervention in 12-weeks, 3 times per week sessions.
  Other Names: Split-belt has two seprate belts.
  Arms: Split-belt

SUMMARY:
Innovative advances in rehabilitation technology have created a split-belt treadmill capable of providing a much needed intervention aimed at limiting mobility disability. When desynchronized, the split-belt treadmill imposes demands on each leg such that the central nervous system must adapt to the challenge. Based on preliminary data from our lab utilizing the split-belt treadmill, the investigators hypothesize this intervention can challenge the locomotor processes required for safe, efficient gait while concurrently providing an aerobic stimulus will produce favorable changes in physical function in older adults at risk for mobility disability.

DETAILED DESCRIPTION:
For this pilot study the investigators will enroll 20 sedentary older adults at risk for disability (usual gait speed ≤ 1.0 m/s). Participants will be assigned to one of two 12-week interventions. Therefore the final training pool will consist of 10 split-belt participants and 10 traditional treadmill participants. Aim 1 will test the hypothesis that compared with a traditional treadmill intervention a split-belt treadmill intervention will result in improved mobility, as measure by 400 meter walk time, as well self reported physical function/disability as measured by the Pepper Assessment Tool for Disability. Aim 2 will test the hypothesis that compared with a traditional treadmill intervention a split-belt treadmill intervention will results in improved gait variability. To date, no experimental study has evaluated these propositions in a controlled trial testing the effects of split-belt training in older adults at risk for disability.

ELIGIBILITY:
Inclusion Criteria:

* aged 65 to 89
* walking speed of ≤ 1 m/s
* ≥ 0.033s of stance time variability
* sedentary as defined by spending less than 20 minutes per week in the past month getting regular physical activity

Exclusion Criteria:

* Significant cognitive impairment
* Failure to provide informed consent
* The need of a walker during the 400 meter walk
* Progressive, degenerative neurological disease
* Severe diabetes, requiring use of insulin

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Change in gait speed, as measure by 400 meter walk time, following 12-weeks of intervention | Participants will be evaluated within 1-week prior to begining the intervention and within 1-week following completion of the 12-week intervention
  Participants will be asked to walk at their usual pace, without over exerting. They can stop for up to 1 min for fatigue or other symptoms. A time limit of 15 minutes to perform the test has been established based on the following considerations.

SECONDARY OUTCOMES:
Change in gait variability from pre to post 12-week intervention | Participants will be evaluated within 1-week prior to begining the intervention and within 1-week following completion of the 12-week intervention
  We will test this working hypothesis by examining changes in spatial and temporal characteristics of gait that occur following 12-weeks of split-belt versus traditional treadmill training. Measures of interest will include variability in stance time, step length, stride length, stride time, swing time, and double limb support time directly from the GAITRite.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Hass, Ph.D., Principal Investigator — University of Florida